CLINICAL TRIAL: NCT01329640
Title: Phase II Feasibility Study of Weekly Paclitaxel Plus Weekly Trastuzumab Followed by Weekly Doxorubicin Plus Daily Oral Cyclophosphamide Plus Weekly Trastuzumab for Locally Advanced HER2-Positive Breast Cancer
Brief Title: Feasibility Study of Metronomic Chemotherapy for Locally Advanced Her2- Positive Breast Cancer (TraQ-Me 01)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Fundação Faculdade de Medicina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 17/2010 TraQ-Me 01
Record Dates: First submitted 2010-11-08; First posted 2011-04-06 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Locally Advanced HER2-positive Breast Cancer
Keywords: Metronimic chemotherapy; Locally Advanced HER2-positive Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel, trastuzumab, doxorrubicin, ciclophosphamide (Experimental)
  Interventions: Device: Drug: Paclitaxel; trastuzumab; doxorrubicin; cyclophosphamide

INTERVENTIONS:
Device: Drug: Paclitaxel; trastuzumab; doxorrubicin; cyclophosphamide — 1. Paclitaxel 100mg/m2 once a week for 8 weeks concomitant to trastuzumab 4mg/kg dose attack after 2mg/kg once a week for 8 weeks followed by;
  2. Doxorrubicin 24mg/m2 once a week concomitantly with oral cyclophosphamide 100mg/day (flat dose) concomitantly with trastuzumab 2mg/kg for 9 weeks
  Other Names: Metronomic chemotherapy with trastuzumab

SUMMARY:
The purpose of this study is to evaluate the safety, effectiveness and cost-effectiveness of metronomic chemotherapy combined with trastuzumab as neoadjuvant therapy for locally advanced HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced breast cancer
* T > 2 cm (any N), or any T and positive node(needle biopsy is required if tumor size is less than 2cm)
* Non-metastatic disease confirmed by computerized tomography and bone scan
* HER2 positive by IHC (+++) and/or Fish (+) according to international definitions (ASCO 2007)
* Normal left ventricular ejection fraction (LVEF)
* Indication of preoperative chemotherapy
* multifocal tumors acceptable provided that the largest tumor is Her2-positive
* ECOG 0-1

Exclusion Criteria:

* Another malignancy within the last 5 years (except curatively treated skin carcinoma, in situ cervix carcinoma, in situ ductal carcinoma of the breast, or in situ lobular carcinoma of the breast)
* Clinically significant comorbidities such as cardiovascular diseases, COPD, renal or liver impairment, psychiatric disorders
* LVEF value below institutional limits of normal range
* Detected or suspected distant metastasis
* Neutrophils lower than 1,500/µL, platelets lower than 100,000/µL, hemoglobin lower than 10 g/dL, AST higher than 2.5x upper limit of normal (ULN), total bilirubin higher than ULN, alkaline phosphatase more than 1.5x ULN

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
INCIDENCE OF FEBRILE NEUTROPENIA | 18 weeks
  INCIDENCE OF FEBRILE NEUTROPENIA WITH METRONOMIC SCHEDULE WILL BE NO HIGHER THAN 10%

SECONDARY OUTCOMES:
TUMOR SIZE | From the beginning of treatment until surgery, disease progression or death
  Efficacy will be assessed by:
  1. Tumor measurements using MRI of the Breast
  2. Pathologic complete response
  3. Progression-free survival
  4. Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, São Paulo, Brazil